CLINICAL TRIAL: NCT00301301
Title: A Retrospective Review of Gemcitabine, Methylprednisolone Cisplatin (GEM-P) With or Without Rituximab in Patients With Relapsed/Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: 2656
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Gemcitabine; Cisplatin; Rituximab

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: Gemcitabine
Drug: Cisplatinum
Drug: Rituximab

SUMMARY:
There has been considerable international /national interest in the GEM-P regimen for treatment of patients with relapsed/refractory lymphoma. Currently, there is no accepted standard therapy for these patients. Since the publication of our experience with this regimen (Study with CCR ethics number 1857 closed to recruitment in July 2003:Ng M, Waters J, Cunningham D et al, Br J Cancer 2005;92:1352-7), we have treated relapsed/refractory lymphoma patients with this regimen and would like to undertake a retrospective review of a sub-group of these patients with diffuse large B cell lymphoma (DLBCL).

Patients treated with GEM-P with or without Rituximab prior to March 2005 for refractory/relapsed DLBCL will be included in the analysis. Accrual of eligible patients currently under follow-up will be performed in clinic at the time of next appointment.

All patients accrued will give informed consent for retrospective case note review, after discussion with a study investigator and after receiving a study information sheet. All eligible patients identified from the pharmacy database, and will be consented at the time of the next clinic appointment, if they are agreeable for the retrospective case note review.

ELIGIBILITY:
Inclusion Criteria:

- a) Age over 18 b) Histological diagnosis of diffuse large B cell lymphoma c) Patients who have received Gemcitabine-cisplatin, methylprednisolone (GEM-P) as per standard unit guidelines with or without Rituximab for relapsed/refractory DLBCL.

d) Informed written consent

Exclusion Criteria:

* a) Medical or psychiatric conditions that compromise the patient's ability to give informed consent b) HIV positive or AIDS related lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 39 participants aged over 18 with histological diagnosid of diffuse large B cell lymphoma and written informed consent. Patients who have received Gemcitabine-cisplatin, methylprednisolone (GEM-P) as per standard unit guidelines with or without Rituximab for relapsed/refractory DLBCL.
Sampling Method: Non-Probability Sample
Enrollment: 39

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS trust, Sutton, Surrey, United Kingdom